CLINICAL TRIAL: NCT04693390
Title: Acupuncture Management of Emergence Agitation in Children Undergoing Tonsillectomy: a Randomized Controlled Trial
Brief Title: Acupuncture in Emergency Delirium After Tonsillectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RC 33/2020
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Emergence Delirium
Keywords: Acupuncture; Emergency Delirium; Tonsillectomy
MeSH Terms: conditions — Emergence Delirium | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): The acupuncture will be applied at points LI4, ST36, HT7, in association with auriculotherapy point Master Cerebral, immediately after induction of anesthesia for 20 minutes
  Interventions: Procedure: Acupuncture
- Standard care group (No Intervention): The patients will follow the standard procedure

INTERVENTIONS:
Procedure: Acupuncture — Application of acupuncture
  Arms: Acupuncture

SUMMARY:
Emergence delirium (ED) (also called emergence agitation) can be defined as a "dissociated state of consciousness in which the child is irritable, uncompromising, uncooperative, incoherent and inconsolable crying, moaning, kicking or thrashing".

Tonsillectomy (with or without adenoidectomy) is a routinely performed operation. Emergence agitation is a frequent phenomenon in children recovering from general anesthesia for tonsillectomy, and increases risk of self-injury. It's not unusual for the post-anesthesia care unit (PACU) staff look that a child, who was asleep just minutes before, starts screaming, pulling out his intravenous line, looks like he's about to fall out of his bed. This condition requires sedatives that may cause undesirable side effects. The cause of emergence delirium and the mechanism of agitation following general anesthesia is unknown. Probably the volatile agents work on some pathways, possibly in the locus coeruleus or amygdala, in the setting of a specific neurodevelopmental stage of the brain.

While emergence delirium can be seen into adulthood, its peak incidence is in younger children (2-7 years of age). The incidence of ED is unclear: anywhere from 2-80%, but when confounders like pain, nausea etc. are controlled, the incidence is probably around 20-30%.

Limited data suggest that acupuncture may be a safe, nonpharmacological treatment for the reduction of pain and agitation in term and preterm infants and that may be an alternative method for preventing ED. In particular a prospective, randomized, double-bind controlled study demonstrated a reduction of the ED in many surgeries, after the electrical stimulation of the heart 7 acupuncture site.

Nearly 400 acupuncture points are known on the body surface and they belong to 14 meridians, running along the human body. After the needle peeling, the nervous free terminations release some polypeptid (the most important is the substantia P) and it increases the excitability of the near nervous free terminations which cause vasodilatation. It has a myorelaxant effect, decreases the level for pain tolerance and make stronger the inhibitor effect of descendent fibers, with production of endogenous endorphins. This is the reason why acupuncture is considered valid in prevention and control of ED.

ELIGIBILITY:
Inclusion criteria

1. Children scheduled to undergo tonsillectomy with or without adenoidectomy
2. American Society of Anesthesiologist (ASA) physical status I or II

Exclusion criteria

1. Coagulation disorders (pro-hemorrhagic status)
2. Neurological disorders (development delay)

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Postoperative agitation evaluated with the PAED scale | Within 5 minutes from arrival in the post anesthesia care unit
  Between groups difference in postoperative agitation assessed by the health personnel with the Pediatric Anesthesia Emergence Delirium (PAED) scale. PAED consists of 5 psychometric items describing emergence behavior, with score ranging from 0 to 20. The severity of ED increases with a higher score. Scores ≥10 indicate the presence of ED.

SECONDARY OUTCOMES:
Postoperative agitation evaluated with the PAED scale | 30 minutes after the arrival in the post anesthesia care unit
  Between groups difference in postoperative agitation assessed by the health personnel with PAED scale. PAED consists of 5 psychometric items describing emergence behavior, with score ranging from 0 to 20. The severity of ED increases with a higher score. Scores ≥10 indicate the presence of ED.
Postoperative agitation evaluated with the Watcha Scale | Within 5 minutes from arrival in the post anesthesia care unit
  Between groups difference in postoperative agitation assessed with the Watcha Scale. The Watcha scale is a 4 points scale, describing the behaviour of the patient; a score >2 indicates emergence delirium.
Postoperative agitation evaluated with the Cravero scale | Within 5 minutes from arrival in the post anesthesia care unit
  Between groups difference in postoperative agitation assessed with the Cravero emergence agitation scale, consisting of five steps from obtunded and unresponsive to wild thrashing behaviour requiring restraint. A score of 4 (from crying and difficult to console to wild thrashing) for 5 or more minutes is indicative of emergency delirium.
Postoperative agitation evaluated with the Watcha Scale | 30 minutes after the arrival in the post anesthesia care unit
  Between groups difference in postoperative agitation assessed with the Watcha Scale. The Watcha scale is a 4 points scale, describing the behaviour of the patient; a score >2 indicates emergence delirium.
Postoperative agitation evaluated with the Cravero scale | 30 minutes after the arrival in the post anesthesia care unit
  Between groups difference in postoperative agitation assessed with the Cravero emergence agitation scale, consisting of five steps from obtunded and unresponsive to wild thrashing behaviour requiring restraint. A score of 4 (from crying and difficult to console to wild thrashing) for 5 or more minutes is indicative of emergency delirium.
Pain evaluated with the FLACC scale | Within 5 minutes from arrival in the post anesthesia care unit
  Between groups difference in pain, evaluated using the Faces, Legs, Activity, Cry and Consolability (FLACC) scale administered by the health personnel. The FLACC tool assesses changes in five categories of behavior (namely: Face, legs, Activity, Crying and Consolability), rating each one on a scale of 0-2. Ten is the maximum score indicating severe pain and a score <2 generally indicates absence of pain. A FLACC score higher than 4 is considered as indicator of moderate pain.
Pain evaluated with the FLACC scale | 30 minutes after the arrival in the post anesthesia care unit
  Between groups difference in pain, evaluated using the FLACC scale administered by the health personnel. The FLACC tool assesses changes in five categories of behavior (namely: Face, legs, Activity, Crying and Consolability), rating each one on a scale of 0-2. Ten is the maximum score indicating severe pain and a score <2 generally indicates absence of pain. A FLACC score higher than 4 is considered as indicator of moderate pain.
Unintended harm caused by patients agitation | Within 5 minutes from arrival in the post anesthesia care unit
  Between groups difference in harming surgical repair, harming self or caregivers, pulling out IV's draws or tubes
Unintended harm caused by patients agitation | 30 minutes after the arrival in the post anesthesia care unit
  Between groups difference in harming surgical repair, harming self or caregivers, pulling out IV's draws or tubes

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Tisato, MD, Principal Investigator — Institute for Maternal and Child Health IRCCS Burlo Garofolo
Locations (1):
- Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste, Italy